CLINICAL TRIAL: NCT01841788
Title: Evaluation of Experimental and Commercial Air-Activated, Adhesive Backed Heat Patches
Brief Title: Evaluation of Experimental Heat Patch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chattem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2012006
Record Dates: First submitted 2013-04-23; First posted 2013-04-29 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2013-04

CONDITIONS: Effects of Heat; Tolerability; Adhesiveness; Dermal Irritation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Thermal Adhesion Patch (Experimental): Group of subjects wearing the experimental patch for 8 hour study duration
  Interventions: Device: Thermal Adhesion Patch
- Marketed Thermal Adhesion Patch (Active Comparator): Group of subjects wearing comparative predicate device for 8 hour study duration.
  Interventions: Device: Marketed Thermal Adhesion Patch
- Placebo Patch (Placebo Comparator): Group of subjects wearing the placebo patch for 8 hour study duration
  Interventions: Device: Placebo Patch

INTERVENTIONS:
Device: Thermal Adhesion Patch
  Arms: Thermal Adhesion Patch
Device: Marketed Thermal Adhesion Patch
  Other Names: ThermaCare Heat Wraps
  Arms: Marketed Thermal Adhesion Patch
Device: Placebo Patch
  Arms: Placebo Patch

SUMMARY:
A disposable, air-activated, adhesive backed heat patch is being developed to provide temporary relief from minor muscular ache and joint pains associated with overexertion strains and sprains as well as minor pain associated with arthritis. The aim of the study is to determine the safety and tolerability of the patch during normal wear conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 18-70 years of age;
* must be in general good health;
* must have absence of any visible disease that might be confused with a skin reaction to the test material;
* Participant's back region must be free of excessive hair, cuts, tattoos, or other aberrations;
* must understand and sign Informed Consent;
* must be considered dependable and able to follow directions;
* must be willing to restrict their activity for the 8 hour patch wear time so that the patches/thermocouples do not come loose;
* must be willing to wear a pouch containing the thermostat and thermocouple wiring for the entire 8 hour period and to return all study supplies to the site at Visit 3. If the items are not returned subject may be invoiced for the value of the unit;
* must be willing not to use any topical products such as lotions, sunscreens, etc. in the test area while participating on the study;
* must agree to use an adequate means of birth control which include: abstinence, partner vasectomy, Intrauterine Device, hormonal implant devices/injections, regular use of birth control pills, birth control patches or condoms with a spermicidal agent;
* Participants are willing to come in with a CLEAN back;
* Participants who are 55 years of age or older, agree to supply a t-shirt to wear at visit two that can be marked on with a marker.

Exclusion Criteria:

* Participants with known skin sensitivity to adhesion products;
* Participants with any skin abnormality likely to be aggravated by the study material such as dermatological disease or infection, rash, atrophic, fragile, or abnormally dry skin, cuts or abrasions at the treatment site;
* Participants who are pregnant or nursing, oral interview only;
* Participants with diabetes or poor circulation;
* Participants unable to tolerate conditions of protocol;
* Participants viewed by the investigator as not being suitable for the study;
* Participants who have had active skin cancer including basal cell carcinoma, or other cancer within one year;
* Participants who are currently participating in another clinical trial;
* Participants who routinely use anti-inflammatory medications (within 5 days of study start (81mg Aspirin is okay)) or immunosuppressive or antihistamine medications within 3 weeks prior to study start (steroid nose/eye drops are ok);
* Participants who currently use allergy injections;
* Participants with history of severe asthma;
* Participants with active or uncontrolled immunologic disorders i.e. AIDS, HIV positive, systemic lupus erythematosus, rheumatoid arthritis;
* Participants with uncontrolled thyroid disease;
* Participants who have any clinically significant chronic illness which could place the subject at increased risk during participation or result in inappropriate dermal response during the study;
* Participants who have used topical medications at the test sites within the past 14 days;
* Participants who have lower midline abdominal pinnicula which may interfere with heat patch/wrap application or evaluation;
* Participants who have a pacemaker, defibrillator or other implantable medical device;
* Participants who have allergies to latex, polyethylene, polypropylene, nickel, chromium or aluminum.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Irritation Evaluation | 8 hours
  A trained skin grader will apply a predetermined scale to the observed skin reactions in the test areas under light supplied by a 100-watt incandescent blue bulb.

SECONDARY OUTCOMES:
Adhesion Evaluation | 8 Hours
  Adhesion will be evaluated to a predetermined scale when the subjects return for visit 3 after approximately 8 hours of wear time.

OTHER OUTCOMES:
Heat Intensity | 8 hours
  Assessed using thermocouple sensors worn between the patch and subject's skin with readings taken every 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Hogan, MD, Principal Investigator — Radiant Research
Locations (1):
- Radiant Research, Inc., Pinellas Park, Florida, United States

IPD SHARING:
Plan to Share IPD: No